CLINICAL TRIAL: NCT01474109
Title: Prospective, Randomized, Placebo-controlled, Double-blind, Multicenter, Parallel Group Study to Assess the Efficacy, Safety and Tolerability of Macitentan in Patients With Ischemic Digital Ulcers Associated With Systemic Sclerosis
Brief Title: Macitentan for the Treatment of Digital Ulcers in Systemic Sclerosis Patients
Acronym: DUAL-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AC-055C301
Record Dates: First submitted 2011-10-31; First posted 2011-11-18 (Estimated); Results first posted 2015-01-06 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2015-01

CONDITIONS: Systemic Sclerosis; Ulcers
Keywords: systemic sclerosis; digital ulcers
MeSH Terms: conditions — Scleroderma, Systemic; Ulcer; digital ulcers | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- macitentan 3mg (Active Comparator): macitentan 3mg tablet once daily
  Interventions: Drug: macitentan 3mg
- macitentan 10mg (Active Comparator): macitentan 10mg tablet once daily
  Interventions: Drug: macitentan 10mg
- placebo (Placebo Comparator): matching placebo once daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: macitentan 3mg — macitentan 3mg tablet once daily
  Other Names: ACT-064992
  Arms: macitentan 3mg
Drug: macitentan 10mg — macitentan 10mg tablet once daily
  Other Names: ACT-064992
  Arms: macitentan 10mg
Drug: placebo — matching placebo once daily
  Arms: placebo

SUMMARY:
The DUAL-1 study is designed as a multicenter, double-blind two-period study with an initial fixed 16-week Period 1, followed by a Period 2 of variable duration. All patients completing Period 1 will continue on their original randomized treatment into Period 2, until the last randomized patient has completed Period 1.

Patients will be randomized in a 1:1:1 ratio (macitentan 3mg: macitentan 10mg: placebo).

The primary objective is to demonstrate the effect of macitentan on the reduction of the number of new digital ulcers in patients with systemic sclerosis and ongoing digital ulcers.

Other objectives include:

* the evaluation of the efficacy of macitentan on hand functionality and DU burden at Week 16 in SSc patients with ongoing DU disease.
* the evaluation of the safety and tolerability of macitentan in these patients.
* the evaluation of the efficacy of macitentan on time to first DU complication during the entire treatment period.

DETAILED DESCRIPTION:
Recurrent digital ulcers (DU) are a manifestation of vascular disease in patients with systemic sclerosis (SSc), are an important source of morbidity and lead to impaired function in these patients. In this study, we are investigating whether treatment with the endothelin receptor antagonist, macitentan, decreases the development of new digital ulcers in patients with SSc. Macitentan is a highly potent, tissue-targeting dual endothelin receptor antagonist. Through complete blockade of endothelin action, macitentan is expected to protect tissue from the damaging effect of elevated endothelin. This therapy is not approved for the treatment of systemic sclerosis, but the use of an ERA is an attractive approach in combating the structural vascular damage observed in SSc leading to complications such as DUs.

ELIGIBILITY:
Inclusion Criteria :

* Patients ≥ 18 years of age
* Women of childbearing potential must use two reliable methods of contraception
* Diagnosis of SSc according to the classification criteria of the American College of Rheumatology (ACR)
* At least one visible, active ischemic digital ulcers (DU) at baseline
* History of at least one additional recent active ischemic DU

Exclusion Criteria :

* DUs due to condition other than SSc
* Symptomatic Pulmonary arterial hypertension (PAH)
* Body mass index (BMI) < 18 kg/m^2
* Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5 x upper limit of the normal range (ULN)
* Hemoglobin < 75% of the lower limit of the normal range
* Systolic blood pressure < 95 mmHg or diastolic blood pressure < 50 mmHg
* Severe malabsorption; any severe organ failure (e.g., lung, kidney), or any life-threatening condition.
* Females who are pregnant or breastfeeding or plan to do so during the course of this study.
* Substance or alcohol abuse or dependence, or tobacco use at any level.
* Treatment with phosphodiesterase type-5 (PDE5) inhibitors.
* Patients on statins, who have received treatment for less than 3 months prior to Screening or whose treatment has not been stable during this period.
* Patients on vasodilators, who have received treatment for less than 2 weeks prior to Screening or whose treatment has not been stable during this period.
* Treatment with prostanoids within 3 months.
* Treatment with disease modifying agents if present for less than 3 months prior to Screening or whose treatment has not been stable for at least 1 month prior to Screening.
* Treatment with oral corticosteroids (> 10 mg/day of prednisone or equivalent).
* Treatment with ERAs within 3 months.
* Systemic antibiotics to treat infected DU(s) within 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2011-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (77):
- United States (15):
  - University of Arizona Arthritis Center, Tucson, Arizona
  - UCLA Medical School - Rheumatology Division Rehabilitation Center, Los Angeles, California
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Sarasota Arthritis Research Center, Sarasota, Florida
  - Ochsner Medical Center, New Orleans, Louisiana
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Michigan - Scleroderma Program, Ann Arbor, Michigan
  - Michigan State University, Grand Rapids, Michigan
  - University of Medicine & Dentistry of New Jersey, UMDNJ Scleroderma Program, New Brunswick, New Jersey
  - The Center for Rheumatology, Albany, New York
  - Shanahan Rheumatology and Immunotherapy, PLLC, Raleigh, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pittsburgh Department of Rheumatology, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
- Australia (5):
  - Royal Adelaide Hospital, Adelaide
  - Wesley Hospital, Thoracic Department, Auchenflower
  - Royal Prince Alfred Hospital, Camperdown
  - St Vincent's Hospital, Fitzroy
  - Menzies Research Institute, Hobart
- Belarus (3):
  - Gomel Regional Clinical Hospital, Homyel
  - Healthcare Institution "Minsk City Hospital #1", Minsk
  - Healthcare Institution "Minsk Clinical Hospital #9", Minsk
- Bulgaria (3):
  - Multiprofile Hospital for Active Treatment "Sveti Pantaleymon", Pleven
  - MHAT "Kaspela" EOOD Plovdiv - Rheumatology Ward, Plovdiv
  - MHAT "Sv. Ivan Rilski" EAD Sofia - Clinic of Rheumatology, Sofia
- Canada (5):
  - Rheumatology Research Associates, Edmonton, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Joseph's Health Care, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec
- Chile (4):
  - Prosalud, Santiago
  - Private Office Marta Aliste, Santiago
  - Hospital San Juan de Dios, Santiago
  - Centro de Estudios Clinicos V, Viña del Mar
- Colombia (2):
  - Medicity S.A.S., Bucaramanga
  - Servimed E.U., Bucaramanga
- Croatia (6):
  - Klinicki Bolnicki Centar Osijek, Osijek
  - University Hospital Centre Rijeka, Rijeka
  - Klinički bolnički centar Split, Split
  - Klinicka Bolnica "Svety Duh", Zagreb
  - Klinička bolnica Dubrava, Zagreb
  - University Hospital Centre Zagreb, Zagreb
- Czechia (3):
  - Lekarna FN Brno, Brno
  - Faculty Hospital Hradec Králové, Hradec Králové
  - Revmatologický ústav Praha, Prague
- Denmark (2):
  - Bispebjerg Hospital København, Copenhagen
  - Odense Universitetshospital, Odense
- Helsingin yliopistollinen keskussairaala (HYKS), Meilahden kolmiosairaala, Reumatologian klinikka, Helsinki, Finland
- Germany (8):
  - Universitätsmedizin Berlin Medizinische Klinik mit Schwerpunkt Rheumatologie und Klinische Immunologie, Berlin
  - Klinik für Dermatologie und Allergologie der Ruhr-Universität Bochum, Bochum
  - Klinik und Poliklinik für Dermatologie und Venerologie der Universität zu Köln, Cologne
  - Medizinische Universitätsklinik Freiburg, Abt. Rheumatologie und klinische Forschung, Freiburg im Breisgau
  - Asklepios Westklinikum Hamburg Abteilung für Gefäßmedizin, Angiologie und Diabetologie, Hamburg
  - Rheumatologie, klinische Immunologie, Nephrologie Asklepios Rheumazentrum Hamburg Asklepios Klinik Altona, Hamburg
  - Akademie für Gefäßkrankheiten eV., Karlsbad
  - Universitäts-Hautklinik Tübingen, Tübingen
- Hungary (3):
  - Budai Irgalmasrendi Kórház, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - Pécsi Tudományegyetem Klinikai Központ, Reumatológiai és Immunológiai Klinika, Pécs
- India (3):
  - Advance Rheumatology Clinic, Hyderabad
  - Krishna Institute of Medical Sciences, Secunderabad
  - Christian Medical College, Vellore
- Italy (3):
  - Azienda Ospedaliera Careggi, Florence
  - Azienda Ospedaliera Policlinico di Modena, Modena
  - Complesso Integrato Columbus, Rome
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - NZOZ Reumed, Lublin
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - Akademicki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocławiu, Wroclaw
- Russia (3):
  - State Healthcare Institution "Penza Regional Clinical Hospital named after N.N. Burdenko", Penza
  - Vladimir Regional State Institution of Healthcare, "Regional Clinical Hospital", Vladimir
  - State Healthcare Institution "Sverdlovsk Regional Clinical Hospital #1", Yekaterinburg
- Ukraine (4):
  - Dinpropetrovsk Regional Clinical Hospital named after I. Mechnykova, Dnipropetrovsk
  - Municipal Institution of Kyiv Regional Council, Kyiv Regional Clinical Hospital, Kyiv
  - Lviv Regional Clinical Hospital, Lviv
  - Internal disease chair of Ukrainian medical dentist academy based on therapy department of Poltava Poltava City Clinical Hospital #1, Poltava

REFERENCES:
- [Derived] Khanna D, Denton CP, Merkel PA, Krieg T, Le Brun FO, Marr A, Papadakis K, Pope J, Matucci-Cerinic M, Furst DE; DUAL-1 Investigators; DUAL-2 Investigators. Effect of Macitentan on the Development of New Ischemic Digital Ulcers in Patients With Systemic Sclerosis: DUAL-1 and DUAL-2 Randomized Clinical Trials. JAMA. 2016 May 10;315(18):1975-88. doi: 10.1001/jama.2016.5258. PMID 27163986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted at 70 centers in 17 countries. First patient randomized was 11 January 2012 and last patient, last visit was 29 November 2013.
Pre-assignment Details: A screening visit was performed between Day -14 and Day -1 of the study. Of the 327 patients screened for the study, 38 were screen failures.
Period: Period 1: Baseline to Week 16
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Started | 95 | 97 | 97
Completed | 88 | 91 | 95
Not Completed | 7 | 6 | 2
Period: Period 2: Week 16 to End of Study
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Started | 88 | 91 | 95
Completed | 70 | 73 | 83
Not Completed | 18 | 18 | 12

BASELINE CHARACTERISTICS:
Population: Full analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo | Total
Number analyzed (Participants) | 95 | 97 | 97 | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 77 | 84 | 84 | 245
  >=65 years | 18 | 13 | 13 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (14.44) | 51.6 (11.10) | 50.6 (12.12) | 51.2 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 81 | 83 | 248
  Male | 11 | 16 | 14 | 41
Race/Ethnicity, Customized [Number; unit: participants]
  White | 86 | 82 | 88 | 256
  Black or African American | 0 | 3 | 1 | 4
  Asian | 5 | 6 | 4 | 15
  Hispanic | 3 | 4 | 3 | 10
  Other | 1 | 2 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Australia | 10 | 9 | 9 | 28
  Belarus | 3 | 3 | 5 | 11
  Bulgaria | 13 | 16 | 17 | 46
  Canada | 1 | 3 | 2 | 6
  Chile | 6 | 7 | 4 | 17
  Colombia | 0 | 2 | 1 | 3
  Croatia | 3 | 1 | 6 | 10
  Czech Republic | 6 | 3 | 5 | 14
  France | 0 | 0 | 1 | 1
  Germany | 9 | 7 | 11 | 27
  Hungary | 4 | 7 | 3 | 14
  India | 4 | 5 | 4 | 13
  Italy | 3 | 3 | 2 | 8
  Poland | 5 | 3 | 3 | 11
  Russian Federation | 6 | 7 | 8 | 21
  Ukraine | 10 | 5 | 7 | 22
  United States | 12 | 16 | 9 | 37

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of New Digital Ulcers (DUs) up to Week 16
Description: DUs were assessed at each visit starting with the screening visit. Only DUs from the proximal interphalangeal joint (PIP) distally (both on the dorsal and volar surface of the hand, including the digital tip) were recorded. The location of each DU was noted. At each subsequent visit the location of each new DU was noted. DUs that occurred and healed between visits and were reported by patients were not recorded as new DUs. The evaluation was performed by an experienced physician or a trained rater with expertise in the assessment of DUs in systemic sclerosis (SSc). For a given patient, DUs were assessed by the same rater at each visit, whenever possible. Any DU that developed over a previously healed ulcer was recorded as a new DU. Incidence rate is adjusted for 16 weeks of observation, hence is calculated as the number of new DUs/total number of observation days.
Time Frame: Baseline to week 16
Population: Full analysis set
Measure: Number; unit: number of new DUs/observation days
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 95 | 97 | 97
number of new DUs/observation days | 0.9082 | 0.9567 | 0.8115
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.706, negative binomial-2 regression (NB-2); NB-2 estimate of new DUs per patient = 1.103, 95% CI 2-sided [0.663 to 1.834] — The estimated value corresponds to the treatment effect i.e. the ratio between the estimated number of new DUs in Macitentan 3 mg and in Placebo
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.360, negative binomial-2 regression (NB-2); NB-2 estimate of new DUs per patient = 1.268, 95% CI 2-sided [0.763 to 2.106] — The estimated value corresponds to the treatment effect i.e. the ratio between the estimated number of new DUs in Macitentan 10 mg and in Placebo

2. Secondary Outcome: Percentage of Participants Without a New DU Up To Week 16
Description: DUs were assessed at each visit starting with the screening visit. Only DUs from the proximal interphalangeal joint (PIP) distally (both on the dorsal and volar surface of the hand, including the digital tip) were recorded. The location of each DU was noted. At each subsequent visit the location of each new DU was noted. DUs that occurred and healed between visits and were reported by patients were not recorded as new DUs. The evaluation was performed by an experienced physician or a trained rater with expertise in the assessment of DUs in systemic sclerosis (SSc). For a given patient, DUs were assessed by the same rater at each visit, whenever possible. Any DU that developed over a previously healed ulcer was recorded as a new DU. Numbers of patients with no new DU at Week 16 are imputed using the last observation carried forward method.
Time Frame: Baseline to week 16
Population: Modified intent-to-treat set. Eleven patients were excluded from the modified intent-treat set due to protocol violations.
Measure: Number; unit: Percentage of participants
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 92 | 92 | 94
Percentage of participants | 64.1 | 63.0 | 67.0
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.6670, Chi-squared; Odds Ratio (OR) = 0.875, 95% CI 2-sided [0.477 to 1.606]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.5518, Chi-squared; Odds Ratio (OR) = 0.832, 95% CI 2-sided [0.454 to 1.524]

3. Secondary Outcome: Percentage of Participants With at Least One DU Complication
Description: DU complications were defined as any one of the following, resulting from DU worsening: critical ischemic crisis necessitating hospitalization; gangrene, (auto)amputation; failure of conservative management; surgical and chemical sympathectomy, vascular reconstructions, or any unplanned surgery in the management of hand SSc manifestations; use of parenteral prostanoids; use of endothelin-receptor antagonists; class II, III, or IV narcotics or a > 50% increase in the existing dose compared with baseline; initiation of systemic antibiotics for the treatment of infection attributed to DUs.
Time Frame: Up to approximately 90 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 92 | 92 | 94
percentage of participants | 14.1 | 19.6 | 19.1
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.3625, Chi-squared; Odds Ratio (OR) = 0.696, 95% CI 2-sided [0.319 to 1.518]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.9362, Chi-squared; Odds Ratio (OR) = 1.030, 95% CI 2-sided [0.498 to 2.133]

4. Secondary Outcome: Change in Hand Functionality Health Assessment Questionnaire - Disability Index (HAQ-DI) Hand Component From Baseline to Week 16
Description: HAQ-DI assesses functional ability regarding fine movements of the upper extremities, locomotor activities in the lower extremities, and movements of the upper and lower limbs. Responses were extracted from the Scleroderma Health Assessment Questionnaire covering 8 domains of functional disability (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other daily activities). A mean score ranging from 0-3 was calculated for each domain, and a composite score by dividing the summed domain scores by the number of domains. The composite score was interpreted as 0 (no impairment in function) to 3 (maximal impairment of function). Hand functionality was assessed using a composite of 4 domains (dressing and grooming, grip, hygiene, and eating).
Time Frame: Baseline to week 16
Population: Modified intention-to-treat set. Eleven patients were excluded from the modified intent-treat set due to protocol violations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 92 | 92 | 94
units on a scale
  Baseline | 1.3 (0.73) | 1.4 (0.70) | 1.3 (0.68)
  Week 16 | 1.2 (0.79) | 1.2 (0.66) | 1.2 (0.73)
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.863, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.1 to 0.2]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.649, ANCOVA; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.1]

5. Secondary Outcome: Health Assessment Questionnaire - Disability Index (HAQ-DI) Overall Score From Baseline to Week 16
Description: HAQ-DI assesses functional ability regarding fine movements of the upper extremities, locomotor activities in the lower extremities, and movements of the upper and lower limbs. Responses were extracted from the Scleroderma Health Assessment Questionnaire covering 8 domains of functional disability (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other daily activities). A mean score ranging from 0-3 was calculated for each domain, and a composite score by dividing the summed domain scores by the number of domains. The composite score was interpreted as 0 (no impairment in function) to 3 (maximal impairment of function).
Time Frame: Baseline to week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 92 | 92 | 94
units on a scale
  Baseline | 1.1 (0.71) | 1.2 (0.66) | 1.1 (0.62)
  Week 16 | 1.1 (0.73) | 1.1 (0.64) | 1.1 (0.67)
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.456, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.440, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.2 to 0.1]

6. Secondary Outcome: Change in Hand Functionality - Hand Disability in Systemic Sclerosis - Digital Ulcers (HDISS-DU) Score From Baseline to Week 16
Description: Patients were asked to answer 24 questions on the use of the hand(s) affected by DUs over the past 7 days on a 6-point scale from 0 (yes without difficulty) to 5 (impossible). The HDISS-DU score is the arithmetic mean of the valid non-missing items. The scores are interpreted as 1 (better ability in completing activities) to 6 (worst ability in completing activities)
Time Frame: Baseline to week 16
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Number analyzed (Participants) | 92 | 92 | 94
units on a scale
  Baseline | 3.0 (1.15) | 3.0 (1.09) | 3.0 (1.09)
  Week 16 | 2.7 (1.14) | 2.6 (0.99) | 2.7 (1.10)
Statistical Analysis 1: Comparison: Macitentan 3mg vs Placebo; Test type: Superiority or Other; p = 0.464, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 2: Comparison: Macitentan 10mg vs Placebo; Test type: Superiority or Other; p = 0.342, ANCOVA; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1]

ADVERSE EVENTS:
Time Frame: From start of study treatment up to 30 days after treatment discontinuation, up to approximately 90 weeks
Description: Safety analysis set. One patient was excluded in the safety analysis set as they did not receive study drug after randomisation.
Arm/Group | Macitentan 3mg | Macitentan 10mg | Placebo
Serious Adverse Events (participants affected / at risk) | 17/94 | 14/97 | 13/97
Other Adverse Events (participants affected / at risk) | 61/94 | 73/97 | 69/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 3mg (N=94) | Macitentan 10mg (N=97) | Placebo (N=97)
INFECTED SKIN ULCER (Infections and infestations) | 0 | 3 | 1
PNEUMONIA (Infections and infestations) | 2 | 1 | 0
BACTERIAL SEPSIS (Infections and infestations) | 0 | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 0 | 1 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 | 1 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0
GANGRENE (Infections and infestations) | 3 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 1 | 0 | 0
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 1 | 0
PLEUROPERICARDITIS (Cardiac disorders) | 0 | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 2 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 1 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 1 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL FIBROSIS (Cardiac disorders) | 1 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 1 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 3 | 2 | 3
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
SYSTEMIC SCLEROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
SCLERODERMA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0
CHEST PAIN (General disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1 | 0
UTERINE PROLAPSE (Reproductive system and breast disorders) | 0 | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 | 0 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
METASTATIC BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0
NEURALGIA (Nervous system disorders) | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 1 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 0
NEPHROTIC SYNDROME (Renal and urinary disorders) | 0 | 0 | 1
RENAL DISORDER (Renal and urinary disorders) | 0 | 0 | 1
SCLERODERMA RENAL CRISIS (Renal and urinary disorders) | 0 | 0 | 1
PROSTATIC OPERATION (Surgical and medical procedures) | 0 | 0 | 1
GRANULOMATOSIS WITH POLYANGIITIS (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 0 | 0
NECROSIS ISCHAEMIC (Vascular disorders) | 1 | 0 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0 | 0
RAYNAUD'S PHENOMENON (Vascular disorders) | 1 | 0 | 1
EXTREMITY NECROSIS (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macitentan 3mg (N=94) | Macitentan 10mg (N=97) | Placebo (N=97)
HEADACHE (Nervous system disorders) | 14 | 19 | 12
INFECTED SKIN ULCER (Infections and infestations) | 7 | 12 | 11
OEDEMA PERIPHERAL (General disorders) | 7 | 12 | 6
SKIN ULCER (Skin and subcutaneous tissue disorders) | 6 | 8 | 9
ANAEMIA (Blood and lymphatic system disorders) | 4 | 8 | 7
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 7 | 4
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 6 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 6 | 5
DIARRHOEA (Gastrointestinal disorders) | 6 | 5 | 7
DIZZINESS (Nervous system disorders) | 4 | 5 | 2
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 5 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 4 | 7
NAUSEA (Gastrointestinal disorders) | 5 | 4 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 4 | 6
BRONCHITIS (Infections and infestations) | 7 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other